CLINICAL TRIAL: NCT07199933
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial of Diacerein in the Treatment of Metabolic Dysfunction-Associated Steatotic Liver Disease in Adults
Brief Title: Diacerein in the Treatment of Metabolic Dysfunction-Associated Steatotic Liver Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hongyan Wu (Other)
Responsible Party: Sponsor-Investigator, Hongyan Wu, Medical graduate student, Nanjing University of Traditional Chinese Medicine
Organization: Nanjing University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025NL-167-02; SJCX25_0997 (Other: Jiangsu Provincial Department of Education)
Record Dates: First submitted 2025-09-08; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: MAFLD
Keywords: MAFLD; Diacerein
MeSH Terms: interventions — diacerein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diacerein 50 mg Capsule (Experimental): Drug: Diacerein Capsules 50mg. Weeks 1-4: 50 mg/day; Weeks 5-24: 100 mg/day.
  Interventions: Drug: Diacerein 50 mg Capsule
- Placebo 50 mg Capsule (Placebo Comparator): Drug: Placebo 50 mg Capsule. Weeks 1-4: 50 mg/day; Weeks 5-24: 100 mg/day.
  Interventions: Drug: Placebo 50 mg

INTERVENTIONS:
Drug: Diacerein 50 mg Capsule — Drug:Diacerein 50 mg Capsule. Weeks 1-4: 50 mg/day; Weeks 5-24: 100 mg/day.
  Other Names: serial numbers:0106408804979; Shuangcuruiyin Jiaonang
  Arms: Diacerein 50 mg Capsule
Drug: Placebo 50 mg — Drug:Placebo 50 mg Capsule. Weeks 1-4: 50 mg/day; Weeks 5-24: 100 mg/day.
  Arms: Placebo 50 mg Capsule

SUMMARY:
Metabolic dysfunction-associated fatty liver disease (MAFLD) is the most common chronic progressive liver disease in China, posing a significant risk for hepatic decompensation, cardiovascular disease (CVD), chronic kidney disease (CKD), and various malignancies. It severely impacts patient quality of life and life expectancy, creating a substantial socioeconomic burden. Currently, no safe and effective drug exists to reverse MAFLD.

Rhubarb (Dà Huáng), a classic Traditional Chinese Medicine (TCM) herb for liver disorders, has a cold nature, bitter taste, and targets the liver, spleen, stomach, large intestine, and pericardium meridians. Its primary active component, Rhein, demonstrates therapeutic potential by targeting key MAFLD pathological processes-insulin resistance, hepatic steatosis, inflammation, and fibrosis. Supporting this, a previous randomized, double-blind, placebo-controlled trial by our group on diacerein (a Rhein derivative) for simple obesity showed that it not only reduced body weight but also improved liver function, Controlled Attenuation Parameter (CAP), and Liver Stiffness Measurement (LSM).

Therefore, this study will investigate diacerein-a marketed drug metabolized to Rhein in vivo-for MAFLD treatment using a randomized, double-blind, placebo-controlled design. The aim is to generate clinical evidence for diacerein and other Rhein derivatives within an integrative medicine framework, providing an evidence-based rationale for expanding the application of rhubarb in MAFLD management.

DETAILED DESCRIPTION:
1. Rhubarb and Its Derivatives Have a Solid Theoretical Basis for Treating MAFLD Metabolic dysfunction-associated fatty liver disease (MAFLD), a chronic progressive liver disease caused by nutritional excess and insulin resistance in genetically susceptible individuals, is now the most common chronic liver disease in China. Despite widespread recognition of its hazards, effective interventions for MAFLD remain lacking. MAFLD's pathogenesis is diverse, involving intertwined factors like insulin resistance, dyslipidemia, inflammation, and fibrosis, making single-target approaches often inadequate. Furthermore, treatment must be tailored to disease stage, addressing metabolic abnormalities, liver injury, and complications concurrently. This complexity means treatment efficacy heavily depends on healthcare resource availability and patient compliance, frequently leading to suboptimal outcomes.

   Traditional Chinese Medicine (TCM), with its unique multi-target, multi-pathway mechanisms and advantages of being simple, convenient, inexpensive, and effective, offers new strategies for MAFLD. TCM theory attributes MAFLD to dietary irregularities, sedentary habits, phlegm-dampness generation, stagnation transforming into heat, and consequent obstruction of the liver collaterals. Clinical epidemiology suggests internal accumulation of dampness-heat is the primary pathogenesis. Rhubarb (Dà Huáng), with its cold nature and bitter taste, is a classic TCM herb for clearing heat, detoxifying, draining fire, and eliminating dampness. Zhang Yuansu's "Origins of Medicine" from the Jin Dynasty notes four actions of rhubarb: 1) expelling substantial heat, 2) removing dampness from the lower energizer, 3) eliminating the old to bring in the new, and 4) dispersing retained food. Rhubarb often serves as the sovereign herb (君药) in MAFLD formulas. Rhein, a primary active component of rhubarb, has demonstrated pharmacological effects against steatosis, inflammation, and fibrosis, making it a potential candidate drug. Its derivative, diacerein, is deacetylated in the gut to rhein, exerting pharmacological effects. Marketed since 1985 for osteoarthritis due to its anti-inflammatory properties (brand name: Diacerein), diacerein has shown promise in clinical trials by our group and others, improving liver function and steatosis markers in obese and type 2 diabetic patients. As a marketed drug derived from a TCM monomer, diacerein combines the multi-target breadth of TCM with the quantifiable, user-friendly nature of Western medicine, representing a potential strategy against current MAFLD treatment challenges.
2. Solid Experimental Foundation for Diacerein in MAFLD Treatment Current MAFLD management focuses on weight/waist circumference reduction, improving insulin resistance, preventing metabolic syndrome/type 2 diabetes, alleviating steatohepatitis, and reversing fibrosis. Extensive pharmacological studies confirm that diacerein and its lead compound, rhein, simultaneously target liver pathology and metabolic abnormalities, providing a robust experimental basis for this study.

   Diacerein and rhein counteract hepatic steatosis, inflammation, and fibrosis. Tobar et al. reported that diacerein (20mg/kg for 10 days) ameliorated steatosis, insulin resistance, and inflammation in diet-induced obese (DIO) mice. Further studies showed it reduces hepatic lipid deposition and improves liver function by inhibiting NLRP3 inflammasome activation and JNK-mediated oxidative stress/apoptosis. Another study found 10 mg/kg/day diacerein improved cholestasis-induced liver fibrosis in mice via the HMGB1/RAGE/NF-κB/JNK pathway. Similarly, rhein improved liver lipid deposition and inflammatory factors in DIO and KK/H1J diabetic mice, and reduced carbon tetrachloride-induced liver fibrosis in rats. Our group confirmed that rhein's amelioration of hepatic steatosis in DIO mice likely occurs by inhibiting fatty acid synthase (FASN) expression and de novo lipogenesis.

   The weight-loss and metabolic benefits of diacerein/rhein are clear. In DIO mice, diacerein reduced body weight and improved insulin sensitivity/glucose tolerance. These metabolic improvements are also documented in type 1 diabetes and PCOS models. Our research further showed rhein reduces fat mass, body weight, and improves insulin resistance in DIO mice by inhibiting macrophage inflammasome activation and promoting adipose tissue thermogenesis.
3. Previous Clinical Studies Suggest Diacerein's Potential for MAFLD Two independent randomized, double-blind, placebo-controlled trials (RCTs) from our group and others, using hepatic steatosis as an efficacy endpoint, suggest diacerein's potential.

An RCT by Nathalie et al. involving 84 patients with type 2 diabetes and NAFLD found two years of diacerein treatment significantly improved Liver Stiffness Measurement (LSM) via Fibroscan, suggesting anti-fibrotic effects. Our RCT in obese patients showed 14 weeks of diacerein not only reduced weight and waist circumference and improved insulin sensitivity but also significantly decreased LSM, Controlled Attenuation Parameter (CAP), and serum ALT levels, indicating potential benefits for liver steatosis, fibrosis, and function alongside metabolic improvements.

In summary, the TCM monomer derivative diacerein has strong TCM theoretical basis, solid pharmacological foundation, and promising clinical evidence for treating MAFLD. However, its efficacy and safety in MAFLD populations require further investigation. Notably, the aforementioned studies relied on Fibroscan, which can be influenced by factors like subcutaneous fat. Therefore, this study proposes a randomized, double-blind, placebo-controlled clinical trial incorporating proton magnetic resonance spectroscopy (¹H-MRS), the non-invasive gold standard for hepatic fat quantification, to comprehensively and objectively evaluate the efficacy and safety of diacerein for adult MAFLD. This will provide reliable evidence for expanding diacerein's indications and future MAFLD drug development, while offering evidence-based support for using rhubarb-based formulations in MAFLD clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand this study and voluntarily sign the informed consent form; willing to comply with and capable of completing all trial procedures.
* Meet the diagnostic criteria for Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD).
* Age ≥18 and ≤60 years, regardless of gender.

Exclusion Criteria:

* Patients with other diseases that may secondarily cause fatty liver disease, including hepatitis B or C virus infection, α-1 antitrypsin deficiency, Wilson's disease, hemochromatosis, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, or HIV infection.
* Alcohol consumption ≥140 g/week for females or ≥210 g/week for males.
* Patients with current or history of cirrhosis or any prior event of hepatic decompensation (i.e., ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, esophageal varices, and/or hepatorenal syndrome).

  (4) Patients with abnormal vital signs, complete blood count (CBC), renal function, or thyroid function (Alanine Aminotransferase [ALT] >5× upper limit of normal [ULN]; Creatinine [Cr] >ULN; Albumin [ALB] <3.5 g/L; TSH >2× ULN; electrolyte imbalances).
* Patients with severe cardiovascular or cerebrovascular diseases (including uncontrolled hypertension, defined as systolic blood pressure >170 mmHg or diastolic blood pressure >100 mmHg), renal diseases, hematopoietic system diseases, psychiatric disorders, autoimmune diseases, or active cancer.
* Glycated Hemoglobin A1c (HbA1c) >7% (in patients without prior history of diabetes).
* Patients with inflammatory bowel disease, intestinal obstruction or pseudo-obstruction, chronic diarrhea, or unexplained abdominal pain.
* Use of medications related to MASLD within 3 months prior to the study (e.g., metformin, thiazolidinediones, dipeptidyl peptidase-4 inhibitors [DPP-4i], glucagon-like peptide-1 receptor agonists [GLP-1RA], sodium-glucose cotransporter-2 inhibitors [SGLT-2i], S-adenosylmethionine [SAM-e], polyenphosphatidylcholine, glycyrrhizin, bicyclol, reduced glutathione, betaine, fish oil, silymarin, obeticholic acid/ursodeoxycholic acid [OCA/UDCA], phosphodiesterase inhibitors [PDEi], gemfibrozil, vitamin E, long-term antibiotics [>1 week], THR-β agonists [resmetirom], initiation or adjustment of lipid-lowering regimens, corticosteroids, immunosuppressants, or Chinese herbal extracts for MASLD treatment [e.g., hawthorn, cassia seed, salvia, notoginseng, kudzu, alisma], or herbal teas [e.g., Ilex chingiana, Kuding tea, Gynostemma, lotus leaf, Pu-erh tea]). Exclusion applies if any of the above criteria are met.
* History of bariatric surgery within the past 2 years.
* History of allergy to diacerein or anthraquinone derivatives.
* Use of diacerein within the past 3 months.
* Pregnant or lactating women, or those planning pregnancy within the next 6 months.
* Participation in another clinical trial involving investigational drugs or devices.
* Contraindications to conventional MRI (e.g., metal implants).
* Inability to complete the study or comply with its requirements, as determined by the investigator.
* Weight gain or loss >5% within 6 months prior to baseline, or >10% within 12 months prior to screening.
* CAP value ≥248 dB/m on Fibroscan but MRI-PDFF <5%.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Absolute change or relative change in Intrahepatic Lipid Content, by Magnetic resonance imaging-proton density fat fraction(MRI-PDFF). | From enrollment to the end of treatment at 6 months
  Absolute percentage change in intrahepatic lipid content, quantified by MRI-PDFF

SECONDARY OUTCOMES:
CAP（Controlled Attenuation Parameter）、LSM（Liver Stiffness Measurement）、ALT（Alanine Aminotransferase）、AST（Aspartate Aminotransferase）、Agile Score、FAST Score（FibroScan-AST Score） | From enrollment to the end of treatment at 6 Months
  CAP(dB/m) and LSM(kPa) values measured by Fibroscan; ALT（U/L）and AST（U/L）levels from liver function tests; the Agile score calculates based on LSM, CAP, ALT, AST, platelet count, age, sex, and diabetes status; the FAST score derives from LSM, CAP, and AST measurements. Agile Score (range 0-1): A score exceeding the threshold of 0.67 warrants high clinical suspicion for advanced hepatic fibrosis.
  FAST Score (range 0-1):
  FAST Score < 0.35: Indicates a very low probability of the patient having both non-alcoholic steatohepatitis (NASH) and significant fibrosis (NASH + ≥F2).
  0.35 ≤ FAST Score ≤ 0.67: Suggests that a liver biopsy may be necessary to confirm the diagnosis.
  FAST Score > 0.67: Indicates a high likelihood that the patient belongs to a high-risk group with NASH and significant fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yingjie Chen, Study Director — Affiliated Hospital of Nanjing University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: No